CLINICAL TRIAL: NCT06791954
Title: The Efficacy of a Telerehabilitation Pilates Program on Lumbopelvic Muscle Morphology in Patients With Fibromyalgia Syndrome
Brief Title: The Efficacy of a Telerehabilitation Pilates Program in Fibromyalgia Syndrome Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, YASEMİN MİRZA, Research Assistant, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024/5012
Record Dates: First submitted 2025-01-08; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Fibromyalgia Syndrome
Keywords: Fibromyalgia; Pain; Telehealth; Telemedicine
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Telerehabilitation group (Active Comparator): Telerehabilitation group
  Interventions: Other: Exercise
- Control group (Other): Control group
  Interventions: Other: Exercise
- Healthy Control Group (No Intervention): The first results were compared

INTERVENTIONS:
Other: Exercise — Clinical pilates program
  Arms: Control group; Telerehabilitation group

SUMMARY:
The study aims to evaluate the effects of a telerehabilitation-based clinical pilates program in patients with fibromyalgia syndrome. A randomized controlled trial was designed. An online clinical Pilates-based exercise program targeting stability and strength that was conducted for 8 weeks with 2 sessions per week was developed for the telerehabilitation group. The same exercise programs for the control group were provided in brochures.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of FMS at least one year before the study
* Stable general health condition for the past 6 months

Exclusion Criteria:

* Inability to cooperate with measurements
* Regular engagement in exercise

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2024-06-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-11-20 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic assessment | First day (at beginning) and last day (8. weeks)
  A 9 MHz linear probe was utilized to determine the transversus abdominis, external oblique, and internal oblique muscles. For the ultrasonographic evaluation of the lumbar multifidus muscles, subjects were positioned in supine and prone positions. A 1.5-6 MHz convex probe was initially placed in a transverse orientation to cover the L4-L5-S1 anatomical region.
McGill core endurance tests | First day (at beginning) and last day (8. weeks)
  The lumbopelvic stability was conducted using McGill core endurance tests, which included tests for trunk flexion, extension, and right and left lateral flexion endurance.
Fibromyalgia Impact Questionnaire | First day (at beginning) and last day (8. weeks)
  The Fibromyalgia Impact Questionnaire (FIQ) is a measure consisting of 10 items that assess physical function, work status, productivity level, depression, anxiety, sleep, pain, stiffness, fatigue, and overall well-being. Higher scores indicate higher disease activity.
Fatigue Severity Scale | First day (at beginning) and last day (8. weeks)
  Fatigue Severity Scale (FSS) consists of a total of nine items. Each item is scored on a scale from 1 to 7. An increase in the total score indicates a higher level of fatigue severity.
Central Sensitization Inventory Short-Form | First day (at beginning) and last day (8. weeks)
  Central Sensitization Inventory Short Form (CSI-SF) is designed to assess the presence of central sensitization and associated symptoms. The total score ranges from 0 to 36, with higher scores indicating greater severity of central sensitization.
Hospital Anxiety and Depression Scale | First day (at beginning) and last day (8. weeks)
  The Hospital Anxiety and Depression Scale comprises 14 items. Odd-numbered items assess anxiety, while even-numbered items evaluate depression. The lowest possible score for each subscale is 0, and the highest is 21.
Numeric Rating Scale | First day (at beginning) and last day (8. weeks)
  The Pain Numeric Rating Scale is a numerical version of the visual analog scale, where patients are asked to indicate the number that best reflects their pain severity on a scale from 0 to 10.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No